CLINICAL TRIAL: NCT03617978
Title: Impact of Passive Leg Raise on Hemodynamic Effect: A Randomized Crossover Experimental Study
Brief Title: Passive Leg Raise During Cardiopulmonary Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lazarski University (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PLR_2018_UL
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Leg Elevation; Hemodynamic Instability; Cardiopulmonary Resuscitation
Keywords: cardiopulmonary resuscitation; hemodynamic; medical simulation; leg elevation

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will not be able to see the device measuring the hemodynamic parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- None Elevation (Experimental): Participant placed on a flat surface. Study participant connected to the measuring hemodynamic parameters device
  Interventions: Procedure: Hemodynamics parameters
- Elevation angle of 20 degrees (Experimental): Participant placed on a flat surface, lower limbs raised and supported at an angle of 20 degrees. Study participant connected to the measuring hemodynamic parameters device
  Interventions: Procedure: Hemodynamics parameters
- Elevation angle of 30 degrees (Experimental): Participant placed on a flat surface, lower limbs raised and supported at an angle of 30 degrees. Study participant connected to the measuring hemodynamic parameters device
  Interventions: Procedure: Hemodynamics parameters
- Elevation angle of 45 degrees (Experimental): Participant placed on a flat surface, lower limbs raised and supported at an angle of 45 degrees. Study participant connected to the measuring hemodynamic parameters device
  Interventions: Procedure: Hemodynamics parameters

INTERVENTIONS:
Procedure: Hemodynamics parameters — real-time evaluation of cardiac output parameters using the ICON device

SUMMARY:
during cardiopulmonary resuscitation, an important element of the procedure is to achieve optimal organ perfusion. For this purpose, high quality chest compressions is one of the basic elements of the procedure. however, similarly as in the case of hypovolemic shock, elevation of the lower limbs may be helpful. The study is a randomized cross-over study and includes the effect of lower limb elevation on hemodynamic parameters in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* voluntary informed consent

Exclusion Criteria:

* hip injury during the six months preceding the examination
* back pain
* kidney damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Cardiac output - CO | during procedure
  the volume of blood that the heart pumps into blood vessels in one minute. It is the product of the frequency of heart contractions (HR) and stroke volume (SV). The parameter is measured using ICON device

SECONDARY OUTCOMES:
Stroke Volume - SV | during procedure
  the amount of blood pressed through one of the heart chambers into the appropriate arterial reservoir during a single heart contraction. The parameter is measured using ICON device
thoracic fluid content - TFC | during procedure
  It is an indicator of total fluid volume, both intracellular and extracellular. The parameter is measured using ICON device

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Lazarski University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available at the main author